CLINICAL TRIAL: NCT06781268
Title: Impact of Life Kinetic Training on Balance, Agility, Jumping, Proprioception, and Cognitive Function in Preadolescent Recreational Fencing Athletes: a Randomized Controlled Trial
Brief Title: Life Kinetic Training Enhances Physical and Cognitive Skills in Young Fencers
Acronym: LiKT-Fence RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Naval Academy (Other)
Collaborators: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Gerasimos Grivas, Lecturer, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-434
Record Dates: First submitted 2025-01-04; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Children; Life kinetic; Motor skills; Exercise; Physical fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Life Kinetic Training Group (Experimental): Participants in this group engaged in Life Kinetic (LK) exercises twice a week for eight weeks. The training program combined physical and cognitive tasks designed to enhance neuroplasticity, improve balance, agility, jumping performance, proprioception, and cognitive functions. The exercises included activities that stimulated mental and physical coordination, aimed at improving overall athletic and mental performance.
  Interventions: Behavioral: Life Kinetic Training
- Control group (No Intervention): Participants in the control group continued their usual recreational fencing training without additional intervention. To match the exposure of the experimental group, they engaged in structured, low-intensity activities unrelated to the objectives of Life Kinetic Training. These activities included light stretching, basic coordination drills, and non-cognitive motor tasks, conducted at the same frequency and duration as the experimental sessions (twice per week for one hour). These activities were designed to simulate a training environment while lacking the cognitive and motor integration components central to the intervention. At the end of the study, participants were fully debriefed about the nature and purpose of their activities, including the rationale for the placebo-like design, as part of the ethical protocol.

INTERVENTIONS:
Behavioral: Life Kinetic Training — Combination of cognitive and physical exercises aimed at improving neuroplasticity, agility, balance, and cognitive functions.
  Arms: Life Kinetic Training Group

SUMMARY:
The purpose of this study was to examine whether Life Kinetic (LK) exercises could improve balance, agility, jumping performance, proprioception, and cognitive functions in recreationally active preadolescents participating in fencing. It specifically aimed to answer if LK training would lead to significant enhancements in these physical and cognitive attributes compared to a control group.

DETAILED DESCRIPTION:
This study evaluated the effects of Life Kinetic (LK) training on balance, agility, jumping performance, proprioception, and cognitive functions in preadolescent recreational fencers. A total of 22 participants, aged 11.6 ± 1.2 years, were randomly assigned to either the experimental group, which performed LK exercises twice weekly for eight weeks, or the control group, which continued their regular fencing activities. The LK exercises combined physical and cognitive tasks to stimulate neuroplasticity and improve overall athletic and mental performance. Key metrics included agility, vertical jump, star balance, Stroop test, and proprioception assessments.

ELIGIBILITY:
Inclusion Criteria:

* Preadolescents aged between 10 and 12 years. Recreationally active in fencing and registered with the same athletic club. Healthy participants with no chronic illnesses, musculoskeletal injuries, or physical limitations in the last six months.

No use of medication within six months prior to the study. Written informed consent provided by the participants and their parents or guardians.

Exclusion Criteria:

* History of chronic illnesses or conditions that could interfere with physical activity (e.g., asthma, cardiovascular issues).

Any injury or physical limitation in the last six months that could impact performance.

Use of medication that could affect physical or cognitive performance within six months before the study.

Participants outside the specified age range (10-12 years). Lack of parental or participant consent.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-05-12 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Counter Movement Jump Measurement | 8 weeks
  The counter movement jump (CMJ) was assessed utilizing the OptoJump Next system (Microgate, Bolzano, Italy). After a self-administered warm-up session, participants performed 3 trials of the counter-movement jump without arm swings, followed by a one-minute rest period, after which they completed the actual CMJ test. Each participant completed three repetitions of the CMJ without arm swings, and the highest result in centimeters (jumping height) was documented as the primary outcome measure. The OptoJump, a dual-beam optical apparatus, quantifies contact and flight durations during jump sequences (or individual jumps). Flight time (tair) was employed to determine the elevation of the body's center of gravity.
Stroop Color and Word Test | 8 weeks
  A Stroop test comprising three distinct conditions was employed (Scarpina and Tagini, 2017). Each condition featured 60 stimuli, arranged with 6 items per line on a 21.5 × 29 cm sheet of paper. In the initial condition, referred to as the reading condition, participants were required to read words printed in black ink, which included the names of colors such as red, green, blue, and yellow. In the second condition, known as the naming condition, participants were instructed to identify the colors of various rectangles. In the third condition, termed the interference condition, participants were required to name the color of the ink used to print the words, while disregarding the semantic content of the words themselves, as they were incongruent with the ink color (e.g., the word "green" printed in red ink). This condition specifically tested the participants' inhibitory control. Across all conditions, participants were instructed to respond as quickly as possible while minimizing erro
Agility T-test | 8 weeks
  The T-test was conducted as previously described (Semenick, 1990). Four cones were positioned in a T formation, with one cone located 9.14 meters from the starting cone and two additional cones placed 4.57 meters on either side of the second cone. All times were recorded using an electronic timing gate (Fusion Sport Inc.), set at a height of 0.75 meters and spanning 3 meters wide, aligned with the marked starting point. Participants were instructed to sprint forward 9.14 meters from the starting line to the first cone, touching it with their right hand. They then shuffled 4.57 meters to the left to reach the second cone, touching it with their left hand. Subsequently, they shuffled 9.14 meters to the right to the third cone, touching it with their right hand, and shuffled 4.57 meters back to the middle cone, touching it with their left hand. Finally, they backpedaled to the starting line. Timing commenced as participants passed through the timing gates and concluded upon their return
Proprioception Test | 8 weeks
  For the position perception test, the IsoMed-2000 isokinetic testing apparatus was utilized (IsoMed-2000 dynamometer; D & R Ferstl GmbH, Hemau, Germany) as described by Wang et al. (2023). Participants wore headphones and an eye mask to eliminate external auditory and visual influences. They maintained their knee joint in the testing position, allowing the isokinetic device (operating at an angular velocity of 1°/s) to automatically flex and extend to the predetermined angles of 30° and 60°.When the angle returned to 0°, the participant moved to the specified position after the automatic stop of the button movement. The difference between the actual angle and the pre-set angle was recorded. Each angle test was conducted three times to calculate the average value.
Y Balance Test | 8 weeks
  Before screening, participants removed their socks and shoes, watched a brief instructional video on performing the Y Balance Test (YBT), and were allowed 4 to 6 practice trials for each limb in each of the three reach directions. Following the practice trials, we measured the lower extremity length from the inferior border of the anterior superior iliac spine to the inferior border of the medial malleolus. Participants then performed dynamic balance tests on both the right and left lower extremities, reaching in the anterior (ANT), posteromedial (PM), and posterolateral (PL) directions with the contralateral limb. Three successful reaches were recorded, and the maximal reach distance in each direction was used for data analysis. To obtain relative values for each direction for both the right and left limbs, the following formula was applied: Relative (normalized) reach distance (%) = (Absolute reach distance / Limb length) × 100.

SECONDARY OUTCOMES:
Body weight | 8 weeks
  Body weight was measured with participants wearing light underwear, standing, and with a precision of 0.1 kg.
Body height | 8 weeks
  Body height was measured with participants standing upright, feet together, back against the wall, and recorded to the nearest 0.1 cm as the maximum distance from the floor to the highest point on the head.
Leg length | 8 weeks
  Leg length was measured using a tape measure from the anterior superior iliac spine (ASIS) to the medial malleolus. Leg length measurements were taken three times for each limb with the participants in a lying position (Sabharwal and Kumar, 2008).

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Naval Academy, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to ensure the privacy and confidentiality of participants. Additionally, explicit consent for data sharing was not obtained from participants or their guardians during the study, and the ethical approval did not include provisions for sharing individual data externally.

REFERENCES:
- [Derived] Yarayan YE, Keskin K, Celik OB, Guder BC, Kurtipek S, Aslan M, Sogut T, Durhan TA, Alkhamees NH, Sheeha BB, Alghannam AF, Al-Mhanna SB, Grivas GV, Batrakoulis A. Impact of life kinetik training on balance, agility, jumping, proprioception, and cognitive function in preadolescent recreational fencing athletes: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Jun 7;17(1):146. doi: 10.1186/s13102-025-01186-3. PMID 40483500